CLINICAL TRIAL: NCT00503542
Title: Management of Vaginal Complaints: A Pilot Study Within a Practice-Based Research Network
Acronym: VCAT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Matthew R. Anderson, MD, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R03HS016050-01 (AHRQ)
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2007-09

CONDITIONS: Vaginitis
Keywords: Vaginitis; Bacterial Vaginosis; Vaginal trichomoniasis; Vulvovaginal candidiasis
MeSH Terms: conditions — Vaginitis; Vaginosis, Bacterial; Trichomonas Vaginitis; Candidiasis, Vulvovaginal | interventions — terconazole; Fluconazole; Metronidazole; Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients primarily with itching or irritation are treated for candidal vaginitis. Patients primarily with vaginal odor are treated for bacterial vaginosis. Patients who did not fit either of the previous groups are treated for both candidal vaginitis and bacterial vaginosis.
  Interventions: Drug: Terazol or oral fluconazole for candidal vaginitis; Drug: Metronidazole or Clindamycin for Bacterial Vaginosis; Drug: Flagyl for definitively diagnosed vaginal trichomoniasis; Other: Empiric Management
- Control (Active Comparator): Patient are examined and a wet mount is prepared. If a definitive diagnosis is made patient is treated for the condition diagnosed. If no diagnosis is made the clinician has the option of either foregoing treatment (watchful waiting) or following the protocol in the experimental group
  Interventions: Drug: Terazol or oral fluconazole for candidal vaginitis; Drug: Metronidazole or Clindamycin for Bacterial Vaginosis; Drug: Flagyl for definitively diagnosed vaginal trichomoniasis

INTERVENTIONS:
Drug: Terazol or oral fluconazole for candidal vaginitis — Intravaginal terazol qhs x 5 nights; oral fluconazole 150 mg po x 1
Drug: Metronidazole or Clindamycin for Bacterial Vaginosis — Metronidazole 500 mg bid x 5 days; Intravaginal metronidazole bid x 5 days; intravaginal clindamycin
  Other Names: Flagyl; Cleocin
Drug: Flagyl for definitively diagnosed vaginal trichomoniasis — Metronidazole 2 gms po x 1
  Other Names: Flagyl
Other: Empiric Management — In this arm of the study women are treated for vaginal complaints purely on the basis of their symptoms.
  Other Names: Flagyl; Metronidazole; Fluconazole; Diflucan
  Arms: Intervention

SUMMARY:
Many women present in primary care with vaginal complaints. The best way of managing these complaints is unclear. This trial will test two different methods of managing patients with vaginal complaints. This is a pilot trial.

DETAILED DESCRIPTION:
Setting: The study will be carried out at two sites within the New York City Research and Improvement Network (NYC RING) an urban Practice Based Research Network comprising 21 clinical sites. Problem: Vaginal symptoms are the most common reason for outpatient gynecological consultation, yet the management of these symptoms is not well grounded in evidence from primary care. Purpose: To prepare for a randomized clinical trial (RCT) to test whether the current standard of care for evaluating vaginal symptoms (which involves looking for specific pathogens) produces better clinical outcomes than a simpler approach, which treats patients based on their symptoms. Methods: 55 premenopausal non-pregnant adult women presenting with vaginal complaints will be randomized into two groups. Women in Group A will be managed on the basis of presenting complaint without physical examination or office laboratory work. Women in Group B will receive a physical examination and office evaluation looking for trichomonads, candida and bacterial vaginosis. They will be managed according to the clinical and office laboratory findings. Patients will be contacted by phone two weeks after consultation to assess symptom resolution, adverse reaction to drugs, satisfaction with care and treatment experiences. Patients will be screened for infection with gonorrhea and chlamydia using a urine antigen test and for trichomoniasis using vaginal culture. Patients whose tests demonstrate trichomoniasis, chlamydia or gonorrhea or who remain symptomatic at the two-week follow-up call will be re-evaluated promptly. Outcomes: AIM 1: Feasibility: The pilot will assess 1) ability to recruit and retain patients, 2) acceptability of study protocols to subjects and 3) prevalence and detection of important sexually transmitted diseases (STD's). AIM 2: Initial evidence of effectiveness: The pilot will provide data on key planned RCT outcome measurements including 1) treatment success rates (allowing estimation of future sample size), 2) need for reconsultation 3) adverse reactions, 4) medication usage and 5) patient satisfaction. Benefit to public health: This pilot study will lead to a RCT of the management of vaginal complaints in primary care. This RCT may support current practice, reinforcing the need for physical exam and laboratory testing in all patients. On the other hand, the trial may support a more limited approach that avoids a pelvic examination. This could result in substantial savings of health care dollars with equivalent clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be premenopausal, non-pregnant women presenting with a chief complaint of vaginal itch, malodor, discharge, pain, irritation or rash. We will accept patient history of being pre-menopausal as valid.

Exclusion Criteria:

* We will exclude women over 45 who have undergone hysterectomy. We will exclude patients who cannot be reached by phone for follow-up interviews. We will exclude pregnant women because of concerns that the diagnosis and treatment of bacterial vaginosis plays a role in pre-term labor prevention.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Self-reported improvement in symptoms | within 2 weeks

SECONDARY OUTCOMES:
Adverse reactions to treatment. | within two weeks
Incidence of STD's | at time of presentation
Vaginal Complaints Scale | within 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R. Anderson, MD, MSc, Principal Investigator — Montefiore Medical Center
Locations (1):
- Family Health Center, The Bronx, New York, United States